CLINICAL TRIAL: NCT02590081
Title: A Prospective Randomized, Double-Blind Parallel Group Trial To Assess The Efficacy And Safety Of Intravenous Dextrose 5% Solution Compare With Normal Saline (Standard Care) In Rinsing During Haemodialysis In Subjects With End Stage Renal Failure (ESRF) With Respect To Systolic Blood Pressure Control Over 3 Months Period.
Brief Title: Effect of Sodium Rinsing Fluid on Blood Pressure and Interdialytic Weight Change in Hemodialysis Patients
Acronym: NSD5
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Penang Hospital, Malaysia (Other Government)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Ong Loke Meng, doctor, Penang Hospital, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NMRR-14-950-20443
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: End-Stage Kidney Disease; Hemodialysis
Keywords: Normal saline; Destrose 5%; Blood pressure; Interdialytic weight gain; thirst level; End Stage Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline (Active Comparator): Normal saline will be used for wash back procedure at the end of hemodiaysis.
  Interventions: Drug: normal saline
- dextrose 5% (Experimental): Dextrose 5% will be used for wash back procedure at the end of hemodiaysis.
  Interventions: Drug: Dextrose 5%

INTERVENTIONS:
Drug: Dextrose 5%
  Arms: dextrose 5%
Drug: normal saline
  Arms: Normal saline

SUMMARY:
This is a prospective, randomized, double-blind, parallel group trial to assess the efficacy and safety of intravenous dextrose 5% solution compare with normal saline (standard care) in wash back procedure during haemodialysis in patients with end stage renal failure (ESRF) with respect to systolic blood pressure control over 3 months period.

The primary objective is to establish efficacy of 5% dextrose solution compared with normal saline (0.9% sodium chloride solution) with respect to systolic blood pressure control in subjects with end stage renal failure (ESRF) on regular hemodialysis. Secondary objectives include monitoring the change in body weight, thirst level and body fluid volume.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, clinically stable maintenance HD patients on a thrice weekly HD regime.
* Have regular hemodialysisforat least 6 months or more.
* Willing and able to provide written, signed informed consent after the nature of the study has been explained.
* Willing and able to comply with all study procedures.
* Age ≥18 years; Age < 75 years old

Exclusion Criteria:

* Diabetes mellitus, Malignancy, Pregnancy
* Inability or unwillingness to provide written consent.
* Inability or unwillingness to comply with the requirements of the protocol as determined by the investigator.
* Simultaneous participation in another clinical study except observational trials
* Any psychological condition which could interfere with the patient's ability to comply with the study protocol
* Inability to perform a blood pressure measurement on the upper limb
* Scheduled for living donor kidney transplant, change to peritoneal dialysis, home HD or plans to relocate to another center during the study period.
* Life expectancy < 6 months
* Recent acute myocardial infarction, congestive cardiac failure, stroke, angina or ICU admission within last 6 months,
* Planned to migrate/move out of the city
* Alcohol abuse/ drug abuse within last 6 months
* Missed > 2 hemodialysis sessions over 1 month
* Requiring non- cuff catheter for hemodialysis
* Admitted for major infection within the last one month

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure control | Time from week 0 until week 12
  post intervention systolic blood pressure reduction compared to baseline

SECONDARY OUTCOMES:
Interdialytic weight gain | Time from week 0 until week 12
  reduced Interdialytic weight gain in experimental group
thirst level | Time from week 0 and week 12
  Dialysis thirst inventory questionnaire to be administer by patient at baseline (week 0) and end of trial (week 12)
intradialytic event | Time from week 0 until week 12
  Any incident occuring during hemodialysis treatment which needed medical intervention. The event are chills and rigor, chest pain, giddiness, cramps, vomiting, blood loss and hypotension.
adverse events | Time from week 0 until week 12
  All observed or spontaneously reported adverse events occur during the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Loke Meng Ong, FRCP, Principal Investigator — Penang Hospital
Locations (15):
- Malaysia (15):
  - Hospital Sultanah Bahiyah, Alor Setar, Alor Star, Kedah
  - UKM Medical Centre, Cheras, Kuala Lumpur
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - UM Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Tuanku Jaafar, Seremban, Negeri Sembilan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Balik Pulau, Balik Pulau, Pulau Pinang
  - Hospital Bukit Mertajam, Bukit Mertajam, Pulau Pinang
  - Penang Hospital, George Town, Pulau Pinang
  - Hospital Kepala Batas, Kepala Batas, Pulau Pinang
  - Seberang Jaya Hospital, Seberang Jaya, Pulau Pinang
  - Hospital Sungai Bakap, Sungai Bakap, Pulau Pinang
  - Miri Hospital, Miri, Sarawak
  - Selayang Hospital, Selayang Baru Utara, Selangor
  - Hospital Serdang, Serdang, Selangor

REFERENCES:
- [Background] Agarwal R. Epidemiology of interdialytic ambulatory hypertension and the role of volume excess. Am J Nephrol. 2011;34(4):381-90. doi: 10.1159/000331067. Epub 2011 Sep 2. PMID 21893975
- [Background] Brennan JM, Ronan A, Goonewardena S, Blair JE, Hammes M, Shah D, Vasaiwala S, Kirkpatrick JN, Spencer KT. Handcarried ultrasound measurement of the inferior vena cava for assessment of intravascular volume status in the outpatient hemodialysis clinic. Clin J Am Soc Nephrol. 2006 Jul;1(4):749-53. doi: 10.2215/CJN.00310106. Epub 2006 May 24. PMID 17699282